CLINICAL TRIAL: NCT07044700
Title: Non-interventional Study of the Effectiveness and Safety of Jardiance in Patients With Heart Failure (HF) of Reduced Ejection Fraction (HFrEF) Compared to Guideline-recommended Non-SGLT2i Therapy Regimens in China: A Sub-study of the Postmarketing Study of Jardiance Among Patients With Heart Failure in China
Brief Title: Real-world Comparative Effectiveness and Safety of Jardiance in Chinese Patients With Heart Failure of Reduced Ejection Fraction
Status: Not yet recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0291
Record Dates: First submitted 2025-06-24; First posted 2025-07-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure of Reduced Ejection Fraction (HFrEF)
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients initiating Jardiance: Initiation of Jardiance for heart failure of reduced ejection fraction (HFrEF) treatment after the launch of HFrEF indication in China
  Interventions: Drug: Jardiance
- Patients initiating other non-SGLT2i medications (ACEi/ARB/ARNI, beta-blockers, and MRA): Initiation of a different guideline-recommended non-sodium-glucose cotransporter-2 inhibitors (non-SGLT2i) medication class (angiotensin-converting-enzyme inhibitors (ACEi)/angiotensin II receptor blocker (ARB)/angiotensin receptor-neprilysin inhibitor (ARNI), betablockers, and mineralocorticoid receptor antagonist (MRA)) for HFrEF treatment, after the launch of HFrEF indication of Jardiance in China
  Interventions: Drug: non-SGLT2 inhibitors

INTERVENTIONS:
Drug: Jardiance — Jardiance
  Other Names: Empagliflozin
  Groups: Patients initiating Jardiance
Drug: non-SGLT2 inhibitors — non-SGLT2 inhibitors
  Groups: Patients initiating other non-SGLT2i medications (ACEi/ARB/ARNI, beta-blockers, and MRA)

SUMMARY:
This study is to provide the effectiveness and safety evidence in patients with heart failure of reduced ejection fraction (HFrEF) initiating Jardiance in real clinical practice in a larger Chinese population.

The primary objective is to compare the risk of the composite outcome of cardiovascular (CV) death or hospitalisation for heart failure (HHF) in heart failure with reduced ejection fraction (HFrEF) patients initiating Jardiance with propensity score (PS) matched HFrEF patients initiating guideline-recommended non-sodium-glucose cotransporter-2 inhibitors (SGLT2i) medications (angiotensin-converting-enzyme inhibitors (ACEi)/angiotensin II receptor blocker (ARB)/angiotensin receptor-neprilysin inhibitor (ARNI), betablockers, and mineralocorticoid receptor antagonist (MRA)) in China, measured by the hazard ratio of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Has at least 1 diagnosis of Heart Failure with Reduced Ejection Fraction (HFrEF) at baseline during the 6-month look-back period (on or prior to the index date)
* Left Ventricular Ejection Fraction (LVEF) ≤40%
* N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) >125pg/mL or Brain Natriuretic Peptide (BNP)≥35 pg/mL
* New users of Jardiance or guideline-recommended non-Sodium-glucose Cotransporter-2 inhibitors (SGLT2i) medications (Angiotensin-converting-enzyme inhibitors (ACEi)/Angiotensin II Receptor Blocker (ARB)/ Angiotensin Receptor-neprilysin Inhibitor (ARNI), beta-blockers, and Mineralocorticoid Receptor Antagonist (MRA)) for HFrEF, who had not used the respective index drug during the look-back period
* Baseline data during the look-back period or on the index date have been collected
* Body mass index (BMI) <45 kg/m2

Exclusion Criteria:

* Patients treated with any SGLT-2i during the look-back period
* Patients treated with any other SGLT-2i on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with heart failure of reduced ejection fraction (HFrEF) included by the heart failure medical union of the national center for cardiovascular diseases (HFMU-NCCD). In the database, heart failure with reduced ejection fraction (HFrEF) is defined as left ventricular ejection fraction (LVEF) <40%.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from the index date to the first hospitalisation for heart failure (HHF) or cardiovascular (CV) death | From the index date to the end date of each individual's follow-up, up to 3 years

SECONDARY OUTCOMES:
Time from the index date to cardiovascular (CV) death | From the index date to the end date of each individual's follow-up, up to 3 years
Time from the index date to the first hospitalisation for heart failure (HHF) | From the index date to the end date of each individual's follow-up, up to 3 years
Total number of HHFs at 30 days after the index date | At 30 days after the index date
Total number of HHFs at 90 days after the index date | At 90 days after the index date
Total number of HHFs at 1 year after the index date | At 1 year after the index date
Time from the index date to all-cause death | From the index date to the end date of each individual's follow-up, up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital; National Center for Cardiovascular Diseases, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com